CLINICAL TRIAL: NCT03113721
Title: Prospective, Non-interventional, Multi-centre Clinical Study to Assess the Clinical Validity of the HBP Assay to Predict Development of Severe Sepsis in Patients With Suspected Infection Following ED Admission
Brief Title: Assessment of Heparin Binding Protein for the Prediction of Severe Sepsis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Axis Shield Diagnostics Ltd (Industry)
Collaborators: Drexel University (Other); York Hospitals (Other); Jefferson Medical College of Thomas Jefferson University (Other); Vanderbilt University Medical Center (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: PEP-FMHBP-005
Record Dates: First submitted 2017-03-24; First posted 2017-04-13 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Sepsis; Septic Shock; Sepsis With Acute Organ Dysfunction
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this prospective, non-interventional, multi-centre clinical study is to assess the clinical validity of the Heparin Binding Protein (HBP) assay for indicating the presence, or outcome, of severe sepsis (including septic shock), over 72 hours, in patients with suspected infection following emergency department admission.

DETAILED DESCRIPTION:
The primary objective of this study is to use HBP concentration to indicate the presence, or outcome, of severe sepsis (including septic shock) at admission and to predict the outcome of severe sepsis (including septic shock) over 72 hours, in patients with suspected infection following emergency department admission.

The secondary objectives of this study are to separately evaluate the performance of HBP concentration to a) indicate the presence of severe sepsis (including severe sepsis) at admission and b) to predict the outcome of severe sepsis (including septic shock) over 72 hours, in patients with suspected infection following emergency department admission.

Further exploratory objectives include evaluating the use of HBP measurement to indicate the outcome of severe sepsis (including septic shock) in patients with suspected infection 12-24 hours after emergency department admission, to compare the use of HBP to other markers of severe infection and to evaluate whether or not different cut-off values are required for the progression and outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age, suspected infection

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (greater than 18 years) presenting to ED with suspected infection
Sampling Method: Non-Probability Sample
Enrollment: 571 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of plasma levels of HBP to evaluate patients with suspected infection for their risk of developing severe sepsis | 72 hours
  The purpose of this measurement is to assess the clinical validity of plasma levels of HBP for indicating the presence, or outcome, of severe sepsis (including septic shock), over 72 hours, in patients with suspected infection following emergency department admission. The concentration of plasma HBP will be compared to the final clinical outcome of the patient to assess the ability of the HBP level to predict clinical progression.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Corbin, MD, Principal Investigator — Drexel University
Locations (5):
- United States (5):
  - Drexel University, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - York Hospitals, York, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No